CLINICAL TRIAL: NCT01549275
Title: Kaohsiung Medical University Hospital
Brief Title: Primary Cell Culture of Hepatic Tumorous Cells From Routine Fine-needle Aspiration
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 990043
Record Dates: First submitted 2012-02-07; First posted 2012-03-09 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cancer cells and cancer-associated fibroblasts
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this prospective study were to evaluate the successful rate of primary culture of hepatocellular carcinoma cells and cancer-associated fibroblasts from the residual specimens in routine fine-needle aspiration of hepatic tumor and the potential application of this method as an additional tool for personalized treatment of hepatocellular carcinoma patients.

DETAILED DESCRIPTION:
Fine-needle aspiration (FNA) cytology or biopsy of hepatic tumor is frequently applied in the collection of specimens because it is considered safe, efficacious, accurate and cost effective. Our previous study from small number of patients showed that specimens obtained from FNA had potential to be applied for primary culture of cancer cells. This study was to modified our method for primary culture of both hepatocellular carcinoma cells and cancer-associated fibroblasts in patients with tumor measuring larger than or equal to 3cm. All patients received one session of aspiration for the diagnosis of hepatic tumor. The aspirated specimens were applied for both cytologic and pathologic examinations at first. After then, 10 mL 0.9% NaCl was aspirated by the same needle connected with the same syringe and injected into 15 mL sterilized centrifugation tube. If the tube contained visible specimens, these specimens were sent for primary culture.

ELIGIBILITY:
Inclusion Criteria:

* patients had residual aspirated specimens for primary culture.

Exclusion Criteria:

* patients did not have residual aspirated specimens for primary culture.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatic tumor measuring larger than or equal to 3 cm underwent fine-needle aspiration of tumor for diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zu Y Lin, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lin ZY, Chuang WL, Chuang YH, Yu ML, Hsieh MY, Wang LY, Tsai JF. Discordant influence of amphotericin B on epirubicin cytotoxicity in primary hepatic malignant cells collected by a new primary culture technique. J Gastroenterol Hepatol. 2006 Feb;21(2):398-405. doi: 10.1111/j.1440-1746.2005.04026.x. PMID 16509865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2010 to January 2013 in Cancer Center and Division of Hepatobiliary Medicine, Department of Internal Medicine, Kaohsiung Medical University Hospital
Pre-assignment Details: A total of 114 patients signed the inform consents. However, 9 patients were excluded due to negative cytological and pathologic results of malignancy in 4 patients, adenocarcinoma in 2 patients and fungal contamination during the preparation of the specimens in 3 patients.
Groups:
- AJCC TNM Staging < = IIIA HCC Patients: Tumor stage is based on the AJCC (American Joint Committee on Cancer) TNM staging system (2010, 7th edition). 76 patients with JACC TNM staging < = IIIA.
- AJCC TNM Staging > = IIIB HCC Patients: 29 patients belonged to AJCC TNM staging > = IIIB.
Period: Overall Study
Arm/Group | AJCC TNM Staging < = IIIA HCC Patients | AJCC TNM Staging > = IIIB HCC Patients
Started | 76 | 29
Completed | 75 | 29
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- AJCC TNM Staging < = IIIA HCC Patients; AJCC TNM Staging > = IIIB HCC Patients: Tumor stage is based on the AJCC (American Joint Committee on Cancer) TNM staging system (2010, 7th edition)
- Total: Total of all reporting groups
Arm/Group | AJCC TNM Staging < = IIIA HCC Patients | AJCC TNM Staging > = IIIB HCC Patients | Total
Number analyzed (Participants) | 76 | 29 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 18 | 49
  >=65 years | 45 | 11 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (12) | 59.6 (14) | 63.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 62 | 24 | 86

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between the Growth Speeds of the Cultured Cells and the AJCC TNM Stage (7th Eds) at Entering of the Study.
Description: Patients were divided into AJCC TNM staging < = IIIA and > = IIIB two groups. The incidences of patients with rapidly proliferative cultured cells in these two groups were compared. Rapidly proliferative group was defined as (1) growth area of cultured cells at the 28th day of primary culture exceeded two times of the growth area measured at the 14th day, or (2) growth area of cultured cells at the 28th day reached > 70% growth area of the flask. Based on the results from special stain, patients in rapidly proliferative group were further divided into patients with rapid proliferation of HCC cells alone, rapid proliferation of HCC cells with concomitant cancer-associated fibroblasts (CAFs) (HCC + CAFs) and CAFs alone.
Time Frame: 28 days after plating of cells
Population: Comparison the incidence of patients with rapidly proliferative cultured cells between two groups
Measure: Number; unit: participants
Arm/Group | AJCC TNM Staging > = IIIB | AJCC TNM Staging < = IIIA HCC Patients
Number analyzed (Participants) | 29 | 76
participants
  Rapidly proliferative cultured cells | 21 | 29
  Rapid Proliferation of HCC with or without CAFs | 14 | 9
  Rapid Proliferation of CAFs alone | 7 | 20
Statistical Analysis 1: Comparison: AJCC TNM Staging > = IIIB vs AJCC TNM Staging < = IIIA HCC Patients; Null hypothesis: There is no significant difference in the incidence of patients with rapidly proliferative cultured cells between two groups; Test type: Superiority or Other; p < 0.005, Chi-squared; degrees of freedom =1
Statistical Analysis 2: Comparison: AJCC TNM Staging > = IIIB vs AJCC TNM Staging < = IIIA HCC Patients; Null hypothesis: There is no significant difference in the incidence of patients with rapidly proliferative cultured HCC cells with or without concomitant cancer-associated fibroblasts between two groups; Test type: Superiority or Other; p < 0.005, Chi-squared; degrees of freedom = 1
Statistical Analysis 3: Comparison: AJCC TNM Staging > = IIIB vs AJCC TNM Staging < = IIIA HCC Patients; Null hypothesis: There is no significant difference in the incidence of patients with rapidly proliferative cultured cancer-associated fibroblasts alone between two groups; Test type: Superiority or Other; p > 0.1, Chi-squared; degrees of freedom = 1

2. Secondary Outcome: Correlation Between the Growth Speeds of Cultured Cells and Worsening of AJCC TNM Stages or HCC Related Death 6 Months After Plating of Cells
Description: 104 Patients with complete follow-up data were further divided into receiving (1) curative treatment of HCC including operative resection and local ablation therapy, (2) palliative transcatheter arterial chemoembolization (TACE), and (3) supportive treatment.
Time Frame: 6 months after plating of cells
Population: Correlation between the growth speeds of cultured cells and worsening of AJCC TNM stages or HCC related death 6 months after plating of cells
Measure: Number; unit: participants
Groups:
- TNM Staging < = IIIA Patients Receiving Curative Treatment: All patient belonged to Child A classification and BCLC (Barcelona Clinic Liver Cancer classification) degree A (14 patients) or B (8 patients).
- TNM Staging < = IIIA Patients Receiving TACE: All patients belonged to Child A classification and BCLC(Barcelona Clinic Liver Cancer classification) degree A or B.
- TNM Staging < = IIIA Patients Receiving Supportive Treatment: 5 patients belonged to BCLC (Barcelona Clinic Liver Cancer classification) degree B and the other 4 patients belonged to BCLC degree C or D.
- TNM Staging > = IIIB Patients Receiving TACE: All patients belonged to Child A classification and BCLC (Barcelona Clinic Liver Cancer classification) degree C.
- TNM Staging > = IIIB Patients Receiving Supportive Treatment: All patients belonged to BCLC (Barcelona Clinic Liver Cancer classification) degree C or D.
Arm/Group | TNM Staging < = IIIA Patients Receiving Curative Treatment | TNM Staging < = IIIA Patients Receiving TACE | TNM Staging < = IIIA Patients Receiving Supportive Treatment | TNM Staging > = IIIB Patients Receiving TACE | TNM Staging > = IIIB Patients Receiving Supportive Treatment
Number analyzed (Participants) | 22 | 44 | 9 | 13 | 16
participants
  Rapidly proliferative cultured cells | 10 | 15 | 3 | 9 | 12
  Rapid growth and worsening stage or death | 0 | 5 | 3 | 4 | 11
  Slow growth and worsening staging or death | 0 | 2 | 1 | 0 | 2
  Rapid growth of HCC cells and worsening | 0 | 2 | 2 | 4 | 8
Statistical Analysis 1: Comparison: TNM Staging < = IIIA Patients Receiving Curative Treatment; null hypothesis: There is no significant difference in the incidence of change in AJCC TNM stages and survivals 6 months after plating of cells between patients with rapidly and slowly proliferative cultured cells; Test type: Superiority or Other; p = 1, Fisher Exact; degrees of freedom = 1
Statistical Analysis 2: Comparison: TNM Staging < = IIIA Patients Receiving TACE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.032, Fisher Exact; degrees of freedom = 1
Statistical Analysis 3: Comparison: TNM Staging < = IIIA Patients Receiving Supportive Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.048, Fisher Exact; degrees of freedom = 1
Statistical Analysis 4: Comparison: TNM Staging > = IIIB Patients Receiving TACE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.176, Fisher Exact; degrees of freedom = 1
Statistical Analysis 5: Comparison: TNM Staging > = IIIB Patients Receiving TACE; Null hypothesis: There is no significant difference in the incidence of change in AJCC TNM stages and survivals 6 months after plating of cells between patients with rapidly and slowly proliferative HCC cultured cells; Test type: Superiority or Other; p = 0.021, Fisher Exact; degrees of freedom = 1
Statistical Analysis 6: Comparison: TNM Staging > = IIIB Patients Receiving Supportive Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.129, Fisher Exact; degrees of freedom = 1

ADVERSE EVENTS:
Time Frame: This study was carried out from April 2010 to January 2013.
Description: This study was to collect the residual specimens obtained from routine aspiration of hepatic tumor. This process did not have any influence on the participants. Serious and other Adverse Events were not collected/assessed."
Groups:
- HCC Patients Underwent FNA of Tumor: Patients who had residual specimens obtained from ultrasound-guided fine-needle aspiration of hepatic tumor measuring equal or larger than 3cm were included. The residual specimens were applied for primary culture and no additional aspiration of the tumor was performed solely for the collection of specimens for culture. Serious and other Adverse Events were not collected/assessed.
Arm/Group | HCC Patients Underwent FNA of Tumor
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No